CLINICAL TRIAL: NCT04200820
Title: Changing Vertical Self-motion Perception After Trampoline Jumping; Assessing Otolith Function in an Elevator
Brief Title: Changing Vertical Self-motion Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BASEC-Nr: 2019-01759
Record Dates: First submitted 2019-12-09; First posted 2019-12-16 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Vestibular Function Tests
Keywords: Sacculus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trampoline (Experimental): The participants will jump on a mini-trampoline for 30 seconds and then will have a 30 seconds break. This will be repeated 16 times. This resulted in a cumulative total intervention time of 8 minutes.
  Interventions: Diagnostic Test: Trampoline

INTERVENTIONS:
Diagnostic Test: Trampoline — During trampoline training that participants undergo constant change of vestibular stimulation. This triggers deep proprioception as well as other sensory inputs. This trigger might affect strength, body stability, muscle coordinative responses, joint movement amplitudes and spatial integration

SUMMARY:
The objective of this study is to explore the "vertical self-motion perception" on in healthy young individuals using an elevator as accelerator. Secondary aim is to explore the effects of repeated vertical acceleration on vertical vestibular sensibility.

DETAILED DESCRIPTION:
The detection of displacement is important information to maintaining balance, postural control, and gait during daily living activities. This detection of displacement or self-motion perception is accomplished by the human vestibular system, particularly the otolith organs, the sacculus and utriculus. Both primarily respond to whole-body acceleration or tilt in gravity. The saccule and utricle detect linear motion as well as the static orientation of the head relative to gravity, which is itself a linear acceleration. The saccule is more sensitive to vertical acceleration (sensing elevator acceleration) and the utricle is more sensitive to horizontal acceleration (sensing a car accelerate). The signals from the vestibular system are transmitted o the central nervous system for further processing.

Testing the otolith function is difficult since it always a combination of the tested inertial acceleration (t) and gravity (g). Therefore the Vector of acceleration is skew. An isolated vertical direction testing of the saccule is to our knowledge not done. Testing the function of the saccule in an elevator would eliminate the any horizontal accelerations other than gravity. Using the decelerations phase of an elevator ride during both up and down ride could give important inside of the self-motion perception (sensation of acceleration of a subject). The reaction force F which accts on the otolith would be maximal when the elevator ride downwards would stop. The force acting on the otolith when the elevator got upwards is breaking is smaller than g.

A better understanding the adaption of the self-motion perception could be beneficial for patients with hypersensitive vestibular functioning, e.g. patients with vestibular migraine. We hypothesized that (a) healthy subjects change the self-motion perception after hyper-stimulation with repeated vertical acceleration.

The objective of this study is to explore the "vertical self-motion perception" on in healthy young individuals using an elevator as accelerator. Secondary aim is to explore the effects of repeated vertical acceleration on vertical vestibular sensibility.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults
* Signed informed consent after being informed

Exclusion Criteria:

* Acute pain
* Chronic neck pain
* Undergone Neck surgery
* Any vestibular disorder
* Fear of elevators / claustrophobia
* Dizziness handicap inventory score >30

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Change of Vertical Self-Motion Perception Reaction Time (VSMPT) | Changes from before and after the elevator rides will be assessed. The assessments will be executed one minute before and after the trampoline intervention. One assessment will take 15 minutes.
  The VSMPT reflects the time in which a person's ability to sense vertical acceleration. A Raspberry Pi 3 B+ with an inertial measurement unit (IMU) will measure the vertical acceleration of the elevator's acceleration. The subject will be asked to stop the stopwatch he/she feels acceleration / deceleration of the elevator ride. The reaction time and the duration of acceleration / deceleration will be measured. Data will be collected starting on the ground floor as the elevator travelled up to a stop at the higher floor (12 floors up). Thereafter the down ride will be measured.Five-elevator rides up and five down will be measured.

SECONDARY OUTCOMES:
Self-administered neck mobility assessment tool (S-ROM-Neck) | 5 minutes. At the start of the study and before the first elevator measurements the participants are asked to fill out the questionnaire.
  The S-ROM-Neck questionnaire is a self-administered questionnaire that uses visual analog scales (VAS) to measure pain-free active range of motion (ROM) for all neck movements. The patient is asked to place a mark on a 100 mm line (0 mm = "no movement possible" and 100 mm = "as far as possible"). The total score is the sum of the individual scores (min. score (600) = no restrictions and max. score (0) = total restriction)
Dizziness handicap inventory (DHI) | 5 minutes. At the start of the study and before the first elevator measurements the participants are asked to fill out the questionnaire.
  The DHI is a validated, 25-item-self-report questionnaire to evaluate the self-perceived handicapping effects caused by dizziness. The DHI is categorized in three domains; functional (9 questions, 36 points), emotional (9 questions, 36 points) and physical (7 questions, 28 points). Patients will answer the questions with no (0 points), sometimes (2 points) and yes (4 points). The higher the score, the greater the handicap caused by dizziness.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — University Hospital Zurich, Directorate of Research and Education
Locations (1):
- University Hospital Zurich, Directorate of Research and Education, Physiotherapy & Occupational Therapy Research, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Publication